CLINICAL TRIAL: NCT05728736
Title: Acute Effect of Lemborexant on CSF Amyloid-Beta and Tau
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to enrollment difficulties and the inability to obtain necessary study supplies. Five participants signed consent; however, no one was randomized. The study was officially terminated with the funding source on 10/04/2023.
Sponsor: Brendan Lucey (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor-Investigator, Brendan Lucey, Principal Investigator, Sleep Medicine Section Head, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HRPO 202210049
Record Dates: First submitted 2023-02-05; First posted 2023-02-15 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease
Keywords: poor sleep
MeSH Terms: conditions — Alzheimer Disease | interventions — lemborexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- treatment (Experimental): 20 participants will be randomized to take lemborexant 25mg at h.s for two consecutive nights
  Interventions: Drug: Lemborexant 25 mg
- placebo (Placebo Comparator): 10 participants will be randomized to take placebo at h.s. for two consecutive nights.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lemborexant 25 mg — Lemborexant 25mg will be taken nightly for two consecutive nights.
  Other Names: Dayvigo
  Arms: treatment
Drug: Placebo — Placebo will be taken nightly for two consecutive nights
  Other Names: inactive pill; sugar pil
  Arms: placebo

SUMMARY:
This study will look at the effects of lemborexant on Alzheimer's disease biomarkers found in the cerebrospinal fluid (CSF) and blood in individuals who are poor sleepers

DETAILED DESCRIPTION:
This study will determine the acute effect of lemborexant on CNS tau phosphorylation and other Alzheimer's disease biomarkers in individuals with poor sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-80 years
* Any sex
* Any race/ethnicity
* Mini-Mental Status Examination score (MMSE) ≥ 27
* Positive plasma amyloid-beta test (i.e., amyloid-positive)
* Pittsburgh Sleep Quality Index >5

Exclusion Criteria:

* Cognitive impairment as determined by history of MMSE < 27
* Inability to speak or understand English
* Any sleep disorders other than insomnia
* No history of moderate-to-severe sleep-disordered breathing and STOP-Bang score > 5
* History or reported symptoms suggestive of restless legs syndrome, narcolepsy or other sleep disorders
* No more than mild sleep apnea (AHI <16) on PSG
* Sleep schedule outside the range of bedtime 22:00-midnight
* Contraindication to lumbar catheter (anticoagulants; bleeding disorder; allergy to lidocaine or disinfectant; prior central nervous system or lower back surgery)
* Cardiovascular disease requiring medication except for controlled hypertension (PI discretion)
* Stroke
* Hepatic or renal impairment
* Pulmonary disease (PI discretion)
* Type 1 diabetes
* HIV or AIDS
* Neurologic or psychiatric disorder requiring medication (PI discretion)
* Suicidal ideations
* Alcohol, tobacco or marijuana use (PI discretion)
* Use of sedating medications (PI discretion)
* Inability to get out of bed independently
* In the opinion of the investigator, the participant should be excluded due to an abnormal physical examination.
* Current pregnancy
* Body Mass Index >35
* History of migraines (PI discretion)
* History of drug abuse in the last 6 months
* History or presence of any clinically significant medical condition, behavioral or psychiatric disorder (including suicidal ideation), or surgical history based on medical record or patient report that could affect the safety of the subject or interfere with study assessments or in the judgment of the PI participant is not a good candidate.
* Urinary or fecal incontinence
* Concurrently enrolled in another trial of an investigational drug or device

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Change in CNS tau phosphorylation | 48 hours
  Changes in CSF pT181/T181 ratio compared to placebo

SECONDARY OUTCOMES:
Changes in other CSF AD biomarkers | 48 hours
  Changes in CSF pS202/S202, pT217/T217, and amyloid-beta

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Lucey, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT05728736/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT05728736/ICF_001.pdf